CLINICAL TRIAL: NCT04101513
Title: The Natural History of Parkinson's Disease-associated Spinal Disorders
Status: Withdrawn | Type: Observational
Why Stopped: Since this project enrolls early-stage Parkinson's patients we hope to develop a registry style study that will allow us to study the progression of spinal disorders in Parkinson patients more effectively.
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Andrew Grossbach, Associate Attending, Ohio State University
Other Study IDs: 2018H0580
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease; Idiopathic Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective single-institution longitudinal study to access quality of life and serial imaging and biodynamic testing to assess spinal disorders associated with Parkinson's disease patients.

DETAILED DESCRIPTION:
This is a prospective single-institution longitudinal study to access quality of life with PROMIS testing, ODI, NDI, VAS and short form 36 health physical component score. The study will also include serial radiographic assessments and biodynamic force plate and hand dynamometer testing. This study will follow for five years post-consent.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Idiopathic Parkinson Disease Early to mid-disease course (Hoehn and Yahr scale 1-3) Age 18-75

Exclusion Criteria:

* Prior spinal fusion Diagnosis of ankylosing spondylitis, diffuse idiopathic spinal hyperostosis (DISH), or other systemic condition that affects spinal function Inability to consent Current incarceration Presence of other medical condition or neurologic condition that would hinder ability to perform biodynamic testing

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients in their early to mid-disease state. (Hoehn and Yahr scale 1-3) Age 18-75 years
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2025-02-14 (Estimated); Study Completion 2027-02-14 (Estimated)

PRIMARY OUTCOMES:
Natural history of spine disorders in idiopathic Parkinson's disease | Consent to five years
  Natural history of spine disorders in idiopathic Parkinson's disease

SECONDARY OUTCOMES:
Clinical impact of Parkinson's related spinal disorders | Consent to five years
  Clinical impact of Parkinson's related spinal disorders assessed by radiographic imaging and biodynamic testing
Factors associated with the development and progression of Parkinson's related spinal disorders | consent to five years
  Factors associated with the development and progression of Parkinson's related spinal disorders by assessing patients reported outcomes
Parameters for optimal management | consent to five years
  Parameters for optimal management will be assessed by imaging and patient's medical records

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Grossbach, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No